CLINICAL TRIAL: NCT02108028
Title: An Exploratory Study of Voicing My CHOiCES as a Tool for Advanced Care Planning in Young Adults With Cancer and Other Chronic Illnesses
Brief Title: Study of Voicing My CHOiCES as a Tool for Advanced Care Planning in Young Adults With Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140079; 14-C-0079
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-11-21

CONDITIONS: HIV; Cancer; Chronic Granulomatous Disease; Dock 8 Deficiency
Keywords: Advance Care Planning Guide; End of life; Natural History
MeSH Terms: conditions — Neoplasms; Granulomatous Disease, Chronic; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cohort 1A / Initial Young Adults with Children: Young adults who have a child(ren) and are 18-39 years diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site. COMPLETE
- Cohort 1B / Comparison Young Adults with Children: Young adults who have children and are 18- 39 years diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site.
- Cohort 2A / Initial Independent Young Adults: Young adults who live independently and are 18-39 years diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site. COMPLETE
- Cohort 2B / Comparison Independent Young Adults: Young adults who live independently and are 18-39 years diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site.
- Cohort 3A / Initial Young Adults No Children, Not Independent: Young adults with no children, not living independently who are 18-39 diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site. COMPLETE
- Cohort 3B / Comparison Young Adults No Children, Not Independent: Young adults with no children, not living independently who are 18-39 diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site.
- Cohort 4 / Non-patient participants: Family members, friends, or health care providers of patient participant. COMPLETE

SUMMARY:
Background:

- There are very few documents to help young adults living with advanced cancer discuss their concerns and end-of-life preferences. A new document, Voicing My CHOiCES, allows young adults to explain what kind of care they would want if they became unable to communicate or make medical decisions on their own. Researchers want to study if this document is helpful.

Objective:

- To study if Voicing My CHOiCES(TM) can reduce anxiety, improve sense of support, and improve communication about advanced care planning.

Eligibility:

- Adults 18 to 39 years old being treated for cancer.

Design:

* Participants will answer questions about their age, sex, employment, religion, health, and marital status. They will also complete several brief questionnaires:

  1. General Anxiety Short Form
  2. Peace, Equanimity and Acceptance in the Cancer Experience
  3. Functional Assessment of Social Support
  4. Quality of Communication
  5. Prior Communication about Advanced Care Planning
* Then a health care professional will introduce Voicing My CHOiCES . Participants will review the document and comment on parts they find relevant. They will also say if any important items are missing. Participants will complete 3 pages of the document with the assistance of a health care provider. They will be asked for positive and negative observations.
* The second stage of the study will take place about 1 month later. Participants will repeat the brief questionnaires listed above. They will be asked if they shared any of the preferences they described when completing the 3 pages of Voicing My CHOiCES during visit 1 with a family member, friend, or health care provider. Research staff will ask the participant for permission to contact the people they spoke with in order to learn whether their conversations about the document were helpful. They will ask for feedback on how to make Voicing My CHOiCES more helpful.

DETAILED DESCRIPTION:
Background:

Discussing end-of-life (EoL) care is very challenging for young adults (YA) living with a life-threatening disease.

While many helpful documents exist to facilitate EoL conversations with adults, few resources exist to aid YA in understanding and accepting their changing physical, emotional and social needs when treatment is no longer effective.

Between 2007-2011, the Pediatric Oncology Branch (07-C-0085) explored the helpfulness of Five Wishes with adolescents and young adults living with HIV or advanced cancer. This research led to the development of a new advance care planning (ACP) guide, Voicing My CHOiCES (VMC). However, Voicing My CHOiCES has not been empirically examined in its completed form.

Objectives:

To determine the perceived helpfulness of VMC.

To determine whether engaging in advanced care planning using VMC is associated with reduced anxiety, improved social support, increased acceptance of illness, and/or improved communication about ACP with family, friends, and/or health care providers.

To assess the helpfulness of the changes made to the original VMC as compared to the revised VMC document.

Eligibility:

Patient Participants:

Age: 18 through 39 years

Known cancer or other chronic illness and enrolled on an NIH protocol or treated at one of the participating sites.

No prior experience using Voicing My CHOiCES

Participants enrolled to assess the helpfulness of changes made to original VMC must be English speaking.

Patients and family/friend and health care providers must be English or Spanish speaking.

Design:

Each subject will complete a baseline assessment of their anxiety pertaining to advance care planning, quality of social support, acceptance of illness, and quality of communication with family, friends and health care providers. They will be asked to review the advance care planning document, Voicing My CHOiCES , and to comment on each section as to whether it can provide an opportunity to address ACP needs for themselves and for other YA their age living with a serious illness. They will also assess whether revisions are needed to the document.

To obtain the perspectives of different YA, the initial study arm included 200 participants, 27 YA who were living independently, 42 YA who have a child(ren) of their own, and 81 YA who neither lived independently or had child(ren). In addition, up to 50 family/friends and health care providers of the participants participated in the follow up assessment. Arm 2 will include up to 80 participants recruited, at the Clinical Center, The Johns Hopkins Hospital, and Rhode Island Hospital (Lifespan) to compare the original Voicing My CHOiCES to the revised document. A total of up to 280 individuals may participate in this study.

A 1-month pre-post design will be used to assess the utility of the document, anxiety, quality of social support, acceptance of illness, communication about EoL planning, and whether the patient participant has shared any of the work completed in the document with a family member, friend, or health care provider.

If the participant had shared the ACP preferences that were documented in Voicing My CHOiCES with a family member or friend, and had consented for us to contact that person, we will obtain the family member or friend s consent and complete a brief interview assessing the helpfulness and limitations of Voicing My CHOiCES for ACP. If the participant had shared the ACP preferences that were documented in Voicing My CHOiCES with their health care provider and had consented for us to talk with that health care provider, a brief interview assessing the helpfulness and limitations of Voicing My CHOiCES for end-of-life planning and whether any changes in the participants health care was made in response to Voicing My CHOiCES , will be documented.

ELIGIBILITY:
* ELIGIBILITY CRITERIA FOR PATIENT PARTICIPANTS (COHORT 1A, 1B, 2A, 2B, 3A & 3B):

INCLUSION CRITERIA:

* Patients must be between ages: 18 through 39 years
* Patients must be diagnosed with cancer or other chronic illness.
* Patients must give informed consent.
* Patients must have a score of 3 or less on the Eastern Cooperative Oncology Group Performance Status Scale (ECOG PS; Appendix
* Patients must be English or Spanish speaking.

  * Cohorts 1B and 2B must be English speaking only.

EXCLUSION CRITERIA:

* Presence of psychotic symptoms or severe psychological distress, which in the judgment of the Principal or Associate Investigator or consulting psychiatrist would compromise the patient s ability to engage in the intervention or is likely to interfere with the study procedures or results.
* Cognitive impairment which in the judgment of the Principal or Associate Investigatorwould compromise the patient s ability to understand the VMC material or is likely to interfere with the study procedures or results.
* Clinically significant, systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgment of the research team would compromise the patient s ability to tolerate or complete this study.
* Participants who have already completed the Voicing My CHOiCES tool.

ELIGIBILITY CRITERIA FOR NON-PATIENT PARTICPANTS (COHORT 4):

INCLUSION CRITERIA:

* Subject must be greater than or equal to 18 years of age
* Family/friend and/or health care providers must be English or Spanish speaking.
* Family/friend and health care providers must provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between 18-39 must be diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at a participating site. Non-Patient participants must be family/friend and/or health care providers of patients diagnosed with cancer or other chronic illness and enrolled on an NIH protocol or treated at one of the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Perceived helpfulness | 2 months
  To determine whether engaging in advance care planning using VMC is associated with reduced anxiety, improved social support, increased acceptance of illness and/or improved communication about ACP with family, friends and/or health care providers.
Improved outcomes | 2 months
  To determine whether engaging in advanced care planning using VMC is associated with reduced anxiety, improved social support, increased acceptance of illness, and/or improved communication about ACP with family, friends, and/or health care providers.
Feasability | 2 months
  To assess the helpfulness of the changes made to the original VMC as compared to the revised VMC document.

SECONDARY OUTCOMES:
Helpfullness vs living & parental status | 2 months
  To examine the helpfulness of VMC by living status (independent living vs. with family of origin) and parental status.
Feasibility | 2 months
  To assess whether further revisions are needed to VMC for use with YA.
Benefit vs burden | 2 months
  To examine the perceived benefit and burden of completing VMC.

CONTACTS AND LOCATIONS:
Overall Officials: Lori S Wiener, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- United States (9):
  - Children's Hospital of Orange County, Orange, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital at Montefiore, The Bronx, New York
  - Rhode Island Hospital (Lifespan), Providence, Rhode Island
  - Cook Childrens Hospital, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Bleyer A. Older adolescents with cancer in North America deficits in outcome and research. Pediatr Clin North Am. 2002 Oct;49(5):1027-42. doi: 10.1016/s0031-3955(02)00035-4. PMID 12430624
- [Background] Bellizzi KM, Smith A, Schmidt S, Keegan TH, Zebrack B, Lynch CF, Deapen D, Shnorhavorian M, Tompkins BJ, Simon M; Adolescent and Young Adult Health Outcomes and Patient Experience (AYA HOPE) Study Collaborative Group. Positive and negative psychosocial impact of being diagnosed with cancer as an adolescent or young adult. Cancer. 2012 Oct 15;118(20):5155-62. doi: 10.1002/cncr.27512. Epub 2012 Mar 13. PMID 22415815
- [Background] Nilsson ME, Maciejewski PK, Zhang B, Wright AA, Trice ED, Muriel AC, Friedlander RJ, Fasciano KM, Block SD, Prigerson HG. Mental health, treatment preferences, advance care planning, location, and quality of death in advanced cancer patients with dependent children. Cancer. 2009 Jan 15;115(2):399-409. doi: 10.1002/cncr.24002. PMID 19110677
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0079.html